CLINICAL TRIAL: NCT03514225
Title: Metacognitive Therapy for Social Anxiety in Youth: A Systematic Replication Series
Brief Title: Metacognitive Therapy for Social Anxiety in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Adrian Wells, Professor of Clinical and Experimental Psychopathology, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 238314
Record Dates: First submitted 2018-03-19; First posted 2018-05-02 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Social Anxiety Disorder; Social Anxiety; Social Phobia
Keywords: Metacognitive Therapy
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metacognitive Therapy for Social Anxiety (Other): Exact sessional content of the MCT intervention is likely to involve attention training and situational attentional refocussing techniques, verbal reattribution strategies aimed to facilitate a reduction of self-processing strategies and to challenge metacognitive beliefs, and between-session tasks for participants to practice at home.
  Interventions: Other: Metacognitive Therapy for Social Anxiety

INTERVENTIONS:
Other: Metacognitive Therapy for Social Anxiety — The transdiagnostic Metacognitive model posits that psychological disorder stems from the activation of a perseverative thinking style called the CAS (Cognitive Attentional Syndrome). This has 3 key elements: worry/rumination, threat-focussed attention and unhelpful coping behaviours. Each of these elements results in extended cognitive responses to negative thoughts, prolonging negative emotions and maintaining an individual's sense of threat. The CAS arises from an individual's positive and negative metacognitive beliefs (beliefs about cognition). Metacognitive Therapy (MCT) aims to bring the CAS under control by modifying metacognitive beliefs and enabling individuals to develop new reactions to negative thoughts.

SUMMARY:
Social anxiety disorder (SAD) is a fear of social situations that involve interacting with other people. Although it can be very upsetting, there are ways to help people deal with it. This study aims to explore the use of a new treatment called Metacognitive Therapy (MCT) for social anxiety in children and teenagers. MCT is a one-to-one talking therapy which works by changing people's patterns of attention and thinking in social situations. By doing this, people with SAD can begin to feel more confident and less anxious when interacting with others.

Findings suggests that MCT works well when treating adults who have social anxiety. However, this treatment has not yet been used with young people. This study hopes to explore whether MCT can help treat SAD in children and teenagers. This information will help us to plan larger studies in the future.

People who would like to take part in this study will be asked to fill in some questionnaires once a week for at least 2 weeks and return these to the researcher in the post. Following this, they will be offered 8 weekly sessions of MCT at their local Child and Adolescent Mental Health Service. Each session will last for about 1 hour. This will involve talking to a clinician about how they think and feel when in social situations, and filling in some more questionnaires. This will allow us to see how their social anxiety changes week-by-week and whether this has improved by the end of treatment (week 8).

1-months after people have had their last session of MCT, they will be asked to complete and return a final set of questionnaires through the post. This will allow us to get a final measure of their social anxiety and see whether any changes in SAD have been maintained.

Primary Questions:

* Is MCT a feasible and acceptable treatment for social anxiety disorder within a child and adolescent population?
* Is MCT associated with improvements in SAD symptoms and functioning?

Secondary Questions:

* Are benefits associated with MCT replicable across subtypes of social anxiety disorder (general and specific)?
* Are any gains associated with MCT for social anxiety disorder maintained at 1 month follow up?

DETAILED DESCRIPTION:
A systematic case replication series utilising an A-B design with 1-month follow-up will be used within this study to replicate MCT intervention across SAD subtypes. (A = no treatment baseline; B = 8 weekly one-one sessions of MCT). This design was chosen as MCT is a relatively novel approach to SAD, particularly within a child and adolescent population.

Recruitment:

Potential participants will be identified by CAMHS Clinicians during routine clinical practice. If the Anxiety Disorders Interview Schedule-IV Child/Parent Version indicates clinical severity of SAD, individuals will be invited to participate in the full study.

This study aims to recruit 5 participants experiencing social anxiety disorder. Participants who drop out of the study during the baseline phase (i.e. before receiving any sessions of MCT intervention) will be replaced by another eligible participant who will be recruited in their place. However, any participants who drop out during the intervention phase of the study will not be replaced.

Phase 1 (Baseline):

During the initial phase of the study, participants will be asked to complete baseline measures once a week for a minimum of 2 weeks (with at least 3 data-points) until stability of scores is achieved. Stability of scores will be defined as 3 consecutive data points showing an increasing or horizontal trend on the primary outcome measure. If the last data point is decreasing, baseline will be extended until stable trends can be plotted, although if stability of scores is not achieved by 6 weeks (i.e. 6 data points) then intervention will be introduced at this point regardless.

Phase 2 (Intervention):

Participants will be invited to attend 8 weekly sessions of MCT at their local CAMHS. Each session will last approximately 1 hour. Participants will be asked to complete sessional measures to allow for monitoring of SAD symptoms and metacognitive beliefs, as well as measures of treatment acceptability.

Phase 3 (Follow-up):

Follow-up will be conducted between 4-6 weeks after the final treatment session. Participants will be asked to complete and return a final set of measures via the post. This will provide a final measure of SAD symptoms and metacognitions and see whether any benefits of receiving MCT have been maintained.

Phase 4 (Exit Interviews):

Participants will be invited to complete an optional, semi-structured exit interview to gather descriptive level information regarding how they found the intervention. This will examine factors such as which components of the intervention were well received.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet criteria for SAD on the ADIS-IV
* Participants must be aged between 13-17 years old at the time of consent
* SAD must be their primary presenting problem (generalised or specific subtype)
* Participants may or may not be taking medication for a mental health difficulty as long as this remains stable during the study
* Participants may or may not have received previous psychological intervention for SAD as long as this is not ongoing

Exclusion Criteria:

* They are aged 18 or above or under the age of 13 at the time of consent
* SAD is not their primary presenting problem
* They are currently undergoing other forms of psychological intervention for SAD or other mental health difficulties [other interventions would need to be suspended for the duration of the study]
* They have a diagnosis of autism spectrum disorder, attention deficit hyperactivity disorder or a learning disability which would impair their ability to participate
* They are non-English speaking
* They are currently demonstrating a high level of risk to themselves or others
* Although participants may also experience low mood, this must not be severe enough to warrant treatment in its own right

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Social Phobia and Anxiety Inventory for Children (SPAI-C; Beidel et al., 1995) | Change in overall SPAI-C score from baseline to 8 weeks post-baseline (end of intervention)
  A 26-item measure of social anxiety, assessing assertiveness, general conversation, physical and cognitive symptoms, avoidance and public performance.

SECONDARY OUTCOMES:
Social Phobia and Anxiety Inventory for Children (SPAI-C; Beidel et al., 1995) | Change in overall SPAI-C score from baseline to 1 month follow-up
  A 26-item measure of social anxiety, assessing assertiveness, general conversation, physical and cognitive symptoms, avoidance and public performance.
Revised Social Phobia Rating Scale (R-SPRS) | Change in R-SPRS scores from baseline to approximately 8 weeks post-baseline (end of intervention)
  A measure of mechanisms (i.e. metacognitive beliefs) which are the focus of modification in MCT, as well as measuring underlying causal processes, self-focussed attention and safety behaviours.
  Item 1 measures distress caused by SAD over the past week on a scale of 0-8. Item 2 measures avoidance over the past week on a scale of 0-8. Item 3 measures self-consciousness over the past week on a scale of 0-8. Item 4 measures safety behaviours, with each listed safety behaviour rated from 0-8. Item 5 measures socially anxious thinking, with each thought rated from 0-100. Item 6 measures worry and rumination over the past week on a scale of 0-8. Item 7 measures threat-monitoring over the past week on a scale of 0-8. Item 8 measures metacognitive beliefs, with each belief rated on a scale of 0-100.
  This scale does not provide an overall score. Each item will be examined individually for change across time as this is a process measure. Higher scores on items indicate worse outcomes.
Revised Social Phobia Rating Scale (R-SPRS) | Change in R-SPRS scores from baseline to 1 month follow-up
  A measure of mechanisms (i.e. metacognitive beliefs) which are the focus of modification in MCT, as well as measuring underlying causal processes, self-focussed attention and safety behaviours.
  Item 1 measures distress caused by SAD over the past week on a scale of 0-8. Item 2 measures avoidance over the past week on a scale of 0-8. Item 3 measures self-consciousness over the past week on a scale of 0-8. Item 4 measures safety behaviours, with each listed safety behaviour rated from 0-8. Item 5 measures socially anxious thinking, with each thought rated from 0-100. Item 6 measures worry and rumination over the past week on a scale of 0-8. Item 7 measures threat-monitoring over the past week on a scale of 0-8. Item 8 measures metacognitive beliefs, with each belief rated on a scale of 0-100.
  This scale does not provide an overall score. Each item will be examined individually for change across time as this is a process measure. Higher scores on items indicate worse outcomes.
Revised Children's Anxiety and Depression Scale (RCADS; Chorpita et al.,2000) | Weekly during baseline, once approximately 8 weeks post-baseline (end of the intervention), and once at 1 month follow-up
  A 47-item screening measure designed to assess selected anxiety and depressive disorders (including SAD).
  Subscales assess:
  Social phobia (9 items; maximum score = 27). Panic disorder (9 items; maximum score = 27). Separation anxiety (7 items; maximum score = 21). Generalised anxiety (6 items; maximum score = 18). Obsessive-compulsive (6 items; maximum score = 18). Major depression (10 items; maximum score = 30).
  In response to each item, participants must select the appropriate response from 'Always' (score = 3), 'Often' (score = 2), 'Sometimes' (score = 1), 'Never' (score = 0).
  Total minimum score = 0. Total maximum score = 141. Higher scores indicate worse outcomes.
Strengths and Difficulties Questionnaire (SDQ; Goodman, 2001) | Weekly during baseline, once approximately 8 weeks post-baseline (end of the intervention), and once at 1 month follow-up
  A 25-item screening questionnaire comprising of 5 scales of 5 items each assessing prosocial behaviour and emotional, conduct, peer relationship and hyperactivity/inattention difficulties.
  Total difficulties score is generated by summing scores from all the scales except the prosocial scale. The resultant score ranges from 0-40. Higher scores indicate worse outcomes.
Session Feedback Questionnaire (SFQ; Evidence Based Practice Unit, 2012) | Intervention session 1 (4-6 weeks after 1st baseline measure, dependent on length of baseline), session 4 (7-10 weeks after 1st baseline measure) and session 8 (11-14 weeks after 1st baseline measure).
  Assesses aspects including whether participants felt listened to and understood session content.
Credibility/Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000) | Intervention session 2 (4-7 weeks after 1st baseline measure, dependent on length of baseline)
  A 6-item self-report measure assessing participant expectancies
Proportion of missed appointments (DNAs) | Proportion of DNAs to be calculated at the end of the intervention phase (11-14 weeks after 1st baseline measure, depending on length of baseline)
  Categorised as when a participant misses an appointment without advance notice
Treatment completion | Proportions to be calculated at the end of the intervention phase of the study (11-14 weeks after 1st baseline measure, depending on length of baseline)
  Completion = when a participant attends all 8 MCT sessions
Drop-out rates | Proportions to be calculated at the end of the intervention phase (11-14 weeks after 1st baseline measure, depending on length of baseline)
  Drop out = when a participant terminates the intervention prior to receiving all 8 sessions

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Wells, Principal Investigator — The University of Manchester
Locations (1):
- Manchester University NHS Foundation Trust (MFT), Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Time Frame: Data will be made available within 12 months of study completion
Access Criteria: Anonymised data will be made available on request (to the Principle Investigator) after publication.

REFERENCES:
- [Background] Beidel, D. C., Turner, S. M. & Fink, C. M. (1996). Assessment of Childhood Social Phobia: Construct, Convergent, and Discriminative Validity of the Social Phobia and Anxiety Inventory for Children (SPAI-C). Psychological Assessment, 8(3), 235-240
- [Background] Wells, A. (2009). Metacognitive Therapy for Anxiety and Depression. New York: Guilford Press
- [Background] Evidence Based Practice Unit (2012). Session Feedback Questionnaire. Retrieved from www.corc.uk.net, 22 September 2017
- [Background] Wells, A., & Matthews, G. (1994). Attention and Emotion: A clinical perspective. Hove UK: Erlbaum.
- [Background] Wells A, Matthews G. Modelling cognition in emotional disorder: the S-REF model. Behav Res Ther. 1996 Nov-Dec;34(11-12):881-8. doi: 10.1016/s0005-7967(96)00050-2. PMID 8990539
- [Background] Wells, A. (1997). Cognitive Therapy of Anxiety Disorders: A Practice Manual and Conceptual Guide. John Wiley & Sons Ltd.
- [Background] Nordahl, H. & Wells, A. (2017). Metacognitive Therapy for Social Anxiety Disorder. Manuscript submitted for publication
- [Background] Silverman, W. K. & Albano, A. M. (1996). The Anxiety Disorders Interview Schedule for Children for DSM-IV: Clinician Manual (Child and Parent Versions). Psychological Corporation, San Antonio, TX
- [Background] Chorpita BF, Yim L, Moffitt C, Umemoto LA, Francis SE. Assessment of symptoms of DSM-IV anxiety and depression in children: a revised child anxiety and depression scale. Behav Res Ther. 2000 Aug;38(8):835-55. doi: 10.1016/s0005-7967(99)00130-8. PMID 10937431
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119